CLINICAL TRIAL: NCT02115113
Title: Multicenter, Prospective, Open-label, Controlled, Randomized, Parallel Groups Study to Evaluate the Renal Function of Adult Liver Transplant Recipients Treated With Two Everolimus-based Immunosuppressive Regimens (Tacrolimus Withdrawal vs. Minimization) Until 12 Months Post-transplant, With a 6-months Follow-up
Brief Title: REnal Function in Liver Transplantation: Everolimus With Calcineurin Inhibitor (CNI)-Sparing sTrategy
Acronym: REFLECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HIT34; 2013-004325-91 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-04-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation, everolimus, CNI-minimization, CNI-elimination, renal function
MeSH Terms: interventions — Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Tacrolimus Elimination Arm) (Experimental): At study start, participants received an Everolimus starting dose of 1.0 mg twice daily in combination with Tacrolimus. Tacrolimus was administered as per center practice. Thereafter, Everolimus doses were adjusted to achieve Everolimus C-0h blood trough levels between 3-8 ng/mL by week 1 after drug initiation until 5 months after transplant. At 5 months after transplant, Everolimus doses were adjusted to achieve C-0h blood trough level target ranges 6-10 ng/mL. Tacrolimus withdrawal was completed by 6 months after transplant.
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Group B (Tacrolimus Minimization Arm) (Active Comparator): At study start, participants received an Everolimus starting dose of 1.0 mg twice daily in combination with Tacrolimus. Tacrolimus was administered as per center practice. Thereafter, Everolimus doses were adjusted to achieve Everolimus C-0h blood trough levels between 3-8 ng/mL by week 1 after drug initiation until 5 months after transplant. At 5 months after transplant, Everolimus doses continued to be adjusted to achieve C-0h blood trough level target ranges 3-8 ng/mL and Tacorlimus doses were adjusted to achieve C-0h blood trough level target ranges 3-5 ng/mL.
  Interventions: Drug: Everolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: Everolimus — Commercial product labeled according to local requirements will be provided as 0.25 mg and 0.75 mg tablets for oral administration.
Drug: Tacrolimus — Commercial product labeled according to local requirements will be provided as 0.5 mg, 1.0 mg and 5.0 mg capsules for oral administration.

SUMMARY:
The purpose of this study was, starting from the Italian clinical practice in liver transplantation, to optimize the immunosuppressive therapy, considering specific patient characteristics as alcoholic cirrhosis, hepatitis C virus (HCV), hepatocellular carcinoma (HCC), and short/long-term implications. Then efficacy and safety of a calcineurin inhibitor (CNI)-withdrawal regimen was evaluated in comparison with a CNI-minimization regimen.

ELIGIBILITY:
Inclusion criteria at Baseline:

* Male and female liver transplant recipients who are ≥ 18 years of age, treated with a tacrolimus-based immunosuppressive regimen, who have received an induction therapy or i.v. steroids as per local clinical practice.
* Recipients of a full-size or technically modified liver allograft will be eligible at 4 weeks (± 7 days) after liver transplantation.
* Allograft is functioning at an acceptable level by the time of Baseline as defined by the AST, ALT, total bilirubin levels ≤ 3 times ULN and INR < 1.5 times ULN.
* Abbreviated MDRD-4 eGFR ≥ 30 mL/min/1.73m2. Serum creatinine results obtained within 5 days prior to Baseline are acceptable.

Inclusion criteria at Randomization:

* Effective tacrolimus minimization, confirmed by stable blood trough levels in the two months prior to randomization, i.e. verification of last two tacrolimus blood trough level ≤ 5 ng/mL in the two months prior to randomization. Investigators should make adjustments in tacrolimus dosing to continue to target trough levels ≤ 5 ng/mL prior to randomization.
* Abbreviated MDRD-4 eGFR ≥ 30 mL/min/1.73m2. Serum creatinine results obtained within 5 days prior to Visit 5 are acceptable.

Exclusion criteria at Baseline:

* Patients who are recipients of multiple solid organ transplants, (e.g., multivisceral or combined liver-kidney transplants), or have previously received an organ or tissue transplanted, or who received an AB0 incompatible transplant.
* Patients who experienced more than one episode of treated biopsy proven acute rejection (BANFF ≥ 3 or RAI ≥ 7) or one steroid-resistant acute rejection.
* Patients who require renal replacement therapy.
* Patients with a confirmed spot urine protein/creatinine ratio that indicates ≥1.0 g/24 hrs of proteinuria.
* History of malignancy of any organ system within the past 5 years whether or not there is evidence of local recurrence or metastases, other than non-metastatic basal or squamous cell carcinoma of the skin or HCC.

Exclusion criteria at Randomization:

* Patients who experienced more than two episodes of treated biopsy proven acute rejection (BANFF ≥ 3 or RAI ≥ 7) since transplantation or one steroid-resistant acute rejection during the run-in period.
* Patients with a confirmed spot urine protein/creatinine ratio that indicates ≥ 3.0 g/24 hrs of proteinuria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Italy (13):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 participants completed run-in but only 50 decided to move forward to randomization.
Pre-assignment Details: This study included a run-in period and a randomization period. Run-in started 4 weeks post-transplant and ended at 5 months post randomization. After run-in, eligible participants were randomized in a 1:1 ratio to tacrolimus elimination or tacrolimus minimization.
Groups:
- Total Enrolled at run-in: Participants, who had a successful liver transplantation and who had initiated a tacrolimus-based regimen and possible induction therapy or intravenous (i.v.) steroids according to local practice, were enrolled into the study 4 weeks (+/- 7 days) after transplantation and started on a everolimus-based regimen with tacrolimus minimization up until 5 months post transplantation.
Period: Participants in Run-in Period
Arm/Group | Group A (Tacrolimus Elimination Arm) | Group B (Tacrolimus Minimization Arm) | Total Enrolled at run-in
Started | 0 | 0 | 78
Completed | 0 | 0 | 68
Not Completed | 0 | 0 | 10
Not completed — Death | 0 | 0 | 1
Not completed — Administrative problems | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3
Period: Participants Randomized
Arm/Group | Group A (Tacrolimus Elimination Arm) | Group B (Tacrolimus Minimization Arm) | Total Enrolled at run-in
Started | 24 | 26 | 0
Completed | 22 | 26 | 0
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Run-in Population: all consented and everolimus-treated patients who entered the run-in treatment period.
  All 78 enrolled patients were included in the run-in treatment period. Treatment started at the randomization period.
Arm/Group | Total Enrolled at run-in
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.73 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Assessed by Estimated Glomerular Filtartion Rate (eGFR)
Description: Renal function was assessed by eGFR using the MDRD-4 formula at 12 months after transplant:
  eGFR = 186.3 * (serum creatinine)-1.154 * age-0.203 * (0.742 for women) * (1.21 if African American) where serum creatinine was in mg/dL and age in years.
Time Frame: At 12 months post-transplant
Population: The safety population, which included all randomized participants who received at least one dose of study medication post-randomization, was considered for the analysis. eGFR values missing at 12 months post transplantation were imputed using the Last Observation carried Forward (LOCF) approach.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Group A (Tacrolimus Elimination Arm) | Group B (Tacrolimus Minimization Arm)
Number analyzed (Participants) | 24 | 26
mL/min/1.73m^2 | 85.50 (3.97) | 80.26 (3.87)
Statistical Analysis 1: Comparison: Group A (Tacrolimus Elimination Arm) vs Group B (Tacrolimus Minimization Arm); Test type: Superiority or Other; p = 0.3013, ANOVA; Mean Difference (Net) = 5.24, 95% CI 2-sided [-4.86 to 15.34], Standard Error of Mean 5.01

2. Secondary Outcome: Percentage of Participants With Treated Biopsy Proven Acute Rejection (tBPAR) Acute Rejection (AR), Graft Loss (GL) or Death (D)
Description: Participants were assessed for tBPAR, AR, GL or death. For all suspected rejection episodes, regardless of initiation of anti-rejection treatment, a liver biopsy was to be performed preferably within 24 hours, latest within 48 hours whenever clinically possible. A treated biopsy proven acute rejection was considered an episode of acute rejection when demonstrated by local pathology reading with a rejection activity index of at least 3 or greater of acute rejection index and when treated with anti-rejection therapy. The allograft was considered lost on the day the subject was re-transplanted or died due to liver failure.
Time Frame: At 12 and 18 months post-transplant
Population: The safety population, which included all randomized participants who received at least one dose of study medication post-randomization, was considered for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tacrolimus Elimination Arm) | Group B (Tacrolimus Minimization Arm)
Number analyzed (Participants) | 24 | 26
Participants
  tBPAR, 12 months | 2 | 1
  AR, 12 months | 2 | 1
  GL, 12 months | 0 | 0
  Death, 12 months | 1 | 0
  tBPAR, 18 months | 2 | 1
  AR, 18 months | 2 | 1
  GL, 18 months | 0 | 0
  Death, 18 months | 1 | 1

3. Secondary Outcome: Change From Baseline (Randomization) in Serum Creatinine at 12 Months Post-transplant
Description: Blood samples were collected to assess serum creatinine.
Time Frame: baseline, 12 months post-transplant
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Group A (Tacrolimus Elimination Arm) | Group B (Tacrolimus Minimization Arm)
Number analyzed (Participants) | 24 | 26
mg/dL | -0.11 (0.04) | -0.05 (0.03)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- Run-in Population Total; Run-in Population Tacrolimus Elimination; Run-in Population Tacrolimus Minimization: At study start, participants received an Everolimus starting dose of 1.0 mg twice daily in combination with Tacrolimus. Tacrolimus was administered as per center practice. Thereafter, Everolimus doses were adjusted to achieve Everolimus C-0h blood trough levels between 3-8 ng/mL by week 1 after drug initiation until 5 months after transplant
- Randomization Treatment Period Tacrolimus Elimination: At 5 months after transplant at randomization, Everolimus doses were adjusted to achieve C-0h blood trough level target ranges 6-10 ng/mL. Tacrolimus withdrawal was completed by 6 months after transplant.
- Randomization Treatment Period Tacrolimus Minimization: At 5 months after transplant at randomization, Everolimus doses continued to be adjusted to achieve C-0h blood trough level target ranges 3-8 ng/mL and Tacorlimus doses were adjusted to achieve C-0h blood trough level target ranges 3-5 ng/mL.
Arm/Group | Run-in Population Total | Run-in Population Tacrolimus Elimination | Run-in Population Tacrolimus Minimization | Randomization Treatment Period Tacrolimus Elimination | Randomization Treatment Period Tacrolimus Minimization
Serious Adverse Events (participants affected / at risk) | 25/78 | 4/24 | 9/26 | 4/24 | 9/26
Other Adverse Events (participants affected / at risk) | 57/78 | 20/24 | 21/26 | 16/24 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Population Total (N=78) | Run-in Population Tacrolimus Elimination (N=24) | Run-in Population Tacrolimus Minimization (N=26) | Randomization Treatment Period Tacrolimus Elimination (N=24) | Randomization Treatment Period Tacrolimus Minimization (N=26)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 2 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2 | 0 | 0 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 2 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 2 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 2 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 6 | 1 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Biliary anastomosis (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Lymphocele (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Population Total (N=78) | Run-in Population Tacrolimus Elimination (N=24) | Run-in Population Tacrolimus Minimization (N=26) | Randomization Treatment Period Tacrolimus Elimination (N=24) | Randomization Treatment Period Tacrolimus Minimization (N=26)
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 3 | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 6 | 0 | 4 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 4 | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 3 | 2 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 7 | 4 | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1 | 5 | 1
Pyrexia (General disorders) | 14 | 4 | 4 | 3 | 4
Cytomegalovirus infection (Infections and infestations) | 4 | 1 | 1 | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 2 | 0 | 2 | 1 | 1
Hepatitis C (Infections and infestations) | 3 | 1 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 1 | 1 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 4 | 0
Blood bilirubin increased (Investigations) | 6 | 2 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 2 | 4 | 2
Transaminases increased (Investigations) | 9 | 4 | 4 | 2 | 2
Weight increased (Investigations) | 2 | 0 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 1 | 4 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 3
Hypercreatininaemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 3 | 1 | 0 | 0
Tremor (Nervous system disorders) | 5 | 2 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 6 | 3 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.